CLINICAL TRIAL: NCT00417040
Title: Collection of Patient-Reported Symptoms and Performance Status Via the Internet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CALGB-70501; CDR0000521898 (Registry Identifier: NCI Physician Data Query); NCI-2009-00489 (Registry Identifier: NCI Clinical Trial Reporting Program); UG1CA189823 (NIH); U10CA037447 (NIH)
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Prostate Cancer; Breast Cancer; Lung Cancer; Colorectal Cancer; Leukemia; Multiple Myeloma
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Breast Neoplasms; Lung Neoplasms; Colorectal Neoplasms; Leukemia; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- (Internet-based STAR database) (Other): Patients are registered into the STAR database, obtain a password, undergo STAR training, and complete a patient-STAR questionnaire after seeing their clinician (baseline self-report) on day 1 of course 2* of chemotherapy. Patients are reminded to complete online STAR questionnaire before seeing their clinician on day 1 of courses 3, 4, 5, and 6* of chemotherapy. Clinicians review these patient reports before creating their own assessment. Patients also complete a patient feedback survey on day 1 of course 4* of chemotherapy. Clinicians complete feedback survey at study completion.
  NOTE: *All time points are based on scheduled therapy with clinical trial CALGB-90401, CALGB-30607, CALGB-30704, CALGB-40601, CALGB-40603, CALGB-40502, CALGB-70604, CALGB-80405, or CALGB-40503.
  Interventions: Other: internet-based intervention; Other: assessment of therapy complications; Other: Questionnaire Administration

INTERVENTIONS:
Other: internet-based intervention — Use the STAR database system
Other: assessment of therapy complications — Use the STAR database system
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This pilot clinical trial studies how well using the internet to collect symptoms and the ability to carry out daily activities works in patients with enrolled on Cancer and Leukemia Group B (CALGB) studies. A study that evaluates a patient's ability to use a clinic waiting room computer to report their symptoms and their ability to carry out daily activities may help doctors understand a patient's use of a computer to report symptoms.

DETAILED DESCRIPTION:
This study enrolled participants who were diagnosed with breast cancer, lung cancer, colorectal cancer, leukemia and multiple myeloma and prostate cancer.

PRIMARY OBJECTIVES:

I. To assess the feasibility of collecting symptom data directly from patients at clinic visits via waiting-area computers.

II. To preliminarily assess the level of agreement between patient and clinician Common Terminology Criteria for Adverse Events (CTCAE) symptom severity scoring, and to measure whether their scores converge when clinicians are exposed to patient self-reports.

OUTLINE:

Patients are registered into the Symptom Tracking and Reporting (STAR) database, obtain a password, undergo STAR training, and complete a patient-STAR questionnaire after seeing their clinician (baseline self-report) on day 1 of course 2* of chemotherapy. Patients are reminded to complete online STAR questionnaire before seeing their clinician on day 1 of courses 3, 4, 5, and 6* of chemotherapy. Clinicians review these patient reports before creating their own assessment. Patients also complete a patient feedback survey on day 1 of course 4* of chemotherapy. Clinicians complete feedback survey at study completion.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Enrolled on clinical trial CALGB-90401, CALGB-30607, CALGB-30704, CALGB-40601, CALGB-40603, CALGB-40502, CALGB-40503, CALGB-70604, or CALGB-80405

PATIENT CHARACTERISTICS:

* Able to read and comprehend English language text
* Able to see a computer screen (i.e., no visual impairments) or be accompanied at visits by someone who can read the screen for the patient

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2006-12 (Actual); Primary Completion 2013-03 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Willingness of approached patients to participate in this study this study | Up to 6 years
Proportion of enrolled patients who submit an online questionnaire at any given follow-up visit any given follow-up visit | Up to 16 weeks
Proportion of total attended visits during the study period at which a questionnaire was completed (completers:visits) which a questionnaire was completed (completers:visits) | Up to 15 weeks

SECONDARY OUTCOMES:
Patient-reported CTCAE symptoms using symptom severity data | At baseline (day 22)
Clinician-reported CTCAE symptoms using symptom severity data clinician reporting at day 43 (when patients report before clinicians; clinicians view those reports) vs at day 22 (patients report symptoms after the clinical encounter) | At baseline (day 22)
Mean severity scores for patient reporting at day 43 | Up to day 43

CONTACTS AND LOCATIONS:
Overall Officials: Ethan Basch, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (95):
- United States (95):
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Valley Medical Oncology Consultants - Castro Valley, Castro Valley, California
  - Valley Medical Oncology, Fremont, California
  - Contra Costa Regional Medical Center, Martinez, California
  - El Camino Hospital Cancer Center, Mountain View, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Breast Surgeons, Incorporated, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Larry G Strieff MD Medical Corporation, Oakland, California
  - Tom K Lee, Incorporated, Oakland, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Doctors Medical Center - San Pablo Campus, San Pablo, California
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - La Grange Memorial Hospital, La Grange, Illinois
  - Center for Cancer Care at OSF Saint Anthony Medical Center, Rockford, Illinois
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Michiana Hematology-Oncology, PC - Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - Michiana Hematology Oncology PC - Plymouth, Plymouth, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC - La Porte, Westville, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Veterans Affairs Medical Center - Iowa City, Iowa City, Iowa
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's Hospital - South, Overland Park, Kansas
  - CCOP - Kansas City, Prairie Village, Kansas
  - CancerCare of Maine at Eastern Maine Medical Center, Bangor, Maine
  - Union Hospital of Cecil County, Elkton, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana-Farber Cancer Institute, Boston, Massachusetts
  - Michiana Hematology Oncology PC - Niles, Niles, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Goldschmidt Cancer Center, Jefferson City, Missouri
  - Truman Medical Center - Hospital Hill, Kansas City, Missouri
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - St. Joseph Medical Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Parvin Radiation Oncology, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Comprehensive Cancer Care, PC, St Louis, Missouri
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - New Hampshire Oncology - Hematology, PA at Payson Center for Cancer Care, Concord, New Hampshire
  - New Hampshire Oncology - Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Lakes Region General Hospital, Laconia, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Norris Cotton Cancer Center at Catholic Medical Center, Manchester, New Hampshire
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Elmhurst Hospital Center, Elmhurst, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - Monter Cancer Center of the North Shore-LIJ Health System, Lake Success, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Don Monti Comprehensive Cancer Center at North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - FirstHealth Moore Regional Community Hospital Comprehensive Cancer Center, Pinehurst, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - Cancer Centers of the Carolinas - Easley, Easley, South Carolina
  - Bon Secours St. Francis Health System, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Faris Road, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Grove Commons, Greenville, South Carolina
  - Greenville Hospital Cancer Center, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Self Regional Cancer Center at Self Regional Medical Center, Greenwood, South Carolina
  - Cancer Centers of the Carolinas - Greer Medical Oncology, Greer, South Carolina
  - Cancer Centers of the Carolinas - Seneca, Seneca, South Carolina
  - Cancer Centers of the Carolinas - Spartanburg, Spartanburg, South Carolina
  - Mountainview Medical, Berlin Corners, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont